CLINICAL TRIAL: NCT06167018
Title: Nurse-administered, Gut-directed Hypnotherapy for Patients With Irritable Bowel Syndrome (IBS).
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Simrén, Proffessor, MD, Sahlgrenska University Hospital
Other Study IDs: 636-12
Record Dates: First submitted 2023-12-01; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurse-delivered, gut-directed hypnotherapy: Adult patients suffering from irritable bowel syndrome (IBS), with symptoms refractory to standard treatment. Patients referred to a tertiary care center were included.
  Interventions: Behavioral: Gut-directed hypnotherapy

INTERVENTIONS:
Behavioral: Gut-directed hypnotherapy — Gut-directed hypnotherapy for patients with irritable bowel syndrome (IBS). Gut-directed hypnotherapy (8-12 sessions), were given either in an individual manner or in a group setting.The hypnosis treatment is administered by two nurses specially trained in Cognitive Behavioral Therapy (CBT) and hypnotherapy. The treatment was based on the North Carolina protocol. Patients assessed gastro-intestinal symptom severity before, during and after treatment, as well as at follow-up.

SUMMARY:
Adult IBS patients with symptoms refractory to standard medical treatment received nurse-administered, gut-directed hypnotherapy. The primary outcome measure was change in gastro-intestinal symptom severity.

DETAILED DESCRIPTION:
IBS patients with symptoms refractory to standard treatment and who were referred to a specialist unit for hypnotherapy, were consecutively included in the study. The patients received gut-directed hypnotherapy given by a nurse trained in Cognitive Behavioral Therapy (CBT) and hypnotherapy. Between 2005 and 2015 patients received 8-12 sessions in an individual manner for 12 weeks. From 2016 the treatment was given in a group format. Effects of treatment were measured by validated questionnaires at baseline and at various time points during the treatment period, as well as after the completion of the treatment at follow-up 6 months, 1 and 2 years after treatment.

ELIGIBILITY:
Inclusion Criteria: IBS diagnosis. -

Exclusion Criteria: Organic GI disease.

-

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult IBS patients with symptoms refractory to standard treatment.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal symptom severity | Baseline (week 0), during treatment (week 6), at treatment completion (week 8), follow-up (6 months, 1 and 2 years after treatment initiation)
  Measured with Irritable Bowel Syndrome- severity scoring system (IBS-SSS). The questionnaire measures severity of GI symptoms and consists of five questions where each score ranges from 0 to 100. A total score of all five questions is calculated ranging from 0 to 500. The higher the score the more severe the GI symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Simrén, Prof, Principal Investigator — Göteborg University
Locations (1):
- Magnus Simrén, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lovdahl J, Blomqvist-Storm M, Palsson OS, Ringstrom G, Tornblom H, Simren M, Trindade IA. Nurse-Administered Gut-Directed Hypnotherapy for Irritable Bowel Syndrome: A Two-Year Follow-Up Study. United European Gastroenterol J. 2025 Sep;13(7):1307-1317. doi: 10.1002/ueg2.70060. Epub 2025 Jun 9. PMID 40491242